CLINICAL TRIAL: NCT00732537
Title: Inhaled Nitric Oxide in Neonates With Elevated A-aDO2 Gradients Not Requiring Mechanical Ventilation
Brief Title: Inhaled Nitric Oxide by Oxygen Hood in Neonates
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Namasivayam Ambalavanan MD and Waldemar A. Carlo MD, Division of Neonatology, Department of Pediatrics, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F990225003
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2008-08

CONDITIONS: Respiratory Failure; Infant; Persistent Fetal Circulation
Keywords: Hypoxia; Respiratory failure; Infant, term; Nitric oxide
MeSH Terms: conditions — Respiratory Insufficiency; Persistent Fetal Circulation Syndrome; Hypoxia | interventions — Nitric Oxide; Oxygen; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inhaled Nitric Oxide (Experimental): iNO started at 20 ppm for 1 hour. The gas was then weaned hourly over the next 4 hours (20 ppm to 10 to 5 to 2.5 to 1 to off).
  Interventions: Drug: inhaled Nitric Oxide
- Placebo (Placebo Comparator): The Oxygen at high concentration (>90%), which was standard therapy for PPHN, was introduced into an oxygen hood (Oxydome ™ disposable hood from Maxtex ® Inc.) using an INOvent (Datex-Ohmeda).
  Interventions: Drug: Oxygen (>90% by hood) - standard therapy

INTERVENTIONS:
Drug: inhaled Nitric Oxide — iNO started at 20 ppm for 1 hour, then weaned hourly over the next 4 hours (20 ppm to 10 to 5 to 2.5 to 1 to off). If >5% drop in oxygen saturation was observed during weaning, study gas was increased to the previous concentration and weaning done 2 hourly. If > 5% drop in oxygen saturation or >5% Methemoglobin was observed during initial administration, the study gas would be weaned over 30 minutes and the infant would exit. The iNO was introduced into an oxygen hood (Oxydome ™ disposable hood from Maxtex ® Inc.) using an INOvent (Datex-Ohmeda). The INOvent ® was connected to the oxyhood by placing the injector module inline on the dry side of the humidifier chamber. Monitoring of O2, NO2, NO was done by placing the end of the sample line inside the oxyhood. A "Masking Shield" covered the Display/Control Panel and Cylinder Gauges, in order to maintain masking of the intervention. Only the respiratory therapist and research coordinator was aware of the allocation assignment.
  Other Names: iNO; Nitric Oxide
  Arms: Inhaled Nitric Oxide
Drug: Oxygen (>90% by hood) - standard therapy — Oxygen (>90% by hood, standard therapy for PPHN prior to intubation) was introduced into an oxygen hood (Oxydome ™ disposable hood from Maxtex ® Inc.) using an INOvent (Datex-Ohmeda). The INOvent ® was connected to the oxyhood by placing the injector module inline on the dry side of the humidifier chamber. If the baby was randomized to the control group and did not receive NO, the INOmax® cylinder was opened and used only to pressurize the system, which prevented the "Low NO Pressure" alarm. A "Masking Shield" covered the Display/Control Panel and Cylinder Gauges, in order to maintain masking of the intervention. Only the respiratory therapist and research coordinator was aware of the allocation assignment.
  Other Names: Oxygen; Head box
  Arms: Placebo

SUMMARY:
Inhaled nitric oxide (iNO) improves oxygenation in term infants with respiratory failure. However, iNO has been primarily used in infants receiving mechanical ventilation. This study is a pilot study to determine if iNO given into an oxygen hood is effective in improving oxygenation in term and near-term infants who have poor oxygenation but who are not yet mechanically ventilated.

DETAILED DESCRIPTION:
Inhaled nitric oxide (iNO) is currently used in the management of ventilated neonates with hypoxemic respiratory failure. We have shown that iNO administered by oxygen hood reduces pulmonary vascular resistance in hypoxia- and group B streptococcus-induced pulmonary hypertension in an animal model (J Perinatol 2002; 22:50-6). Our objective was to determine the feasibility of iNO administration by oxygen hood in neonates with respiratory failure. Methods: A masked randomized controlled trial was performed on eight infants with respiratory failure. Inclusion criteria were: gestation>34 weeks, age<7 days, with post-ductal arterial line, and A-aDO2 400-600 on two consecutive blood gases. Infants were randomized to study gas (iNO at 20 ppm or equivalent flow of O2) for 1 hr which was then weaned over the next 4 hours. The iNO was introduced into an oxygen hood using an INOvent (INO Therapeutics, Inc). The primary outcome was the PaO2 one hour after randomization. Environmental leakage of NO and NO2 were measured. Results: Four infants were randomized to iNO and four to O2 (controls). Two of the four infants given iNO had an increase in PaO2 of >100 mm Hg, while oxygenation was unchanged in the controls. Methemoglobinemia and other adverse effects were not noted in any infant. Environmental levels of NO and NO2 were minimal (<1ppm) to undetectable at >0.3m from the hood. Conclusions: Administration of iNO by oxygen hood is feasible. Larger randomized controlled trials are required to measure the efficacy and determine an appropriate target population for this technique.

ELIGIBILITY:
Inclusion Criteria:

* gestation >34 weeks at birth
* age <7 days
* post-ductal arterial line
* an A-aDO2 of 400 to 600 on two blood gases, at least 30 minutes apart.

Exclusion Criteria:

* Infants with major malformations
* Infants with cardiac disease

Ages: 1 Hour to 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 1999-03; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
PaO2 one hour after the first hour of study gas | one hour after the first hour of study gas

SECONDARY OUTCOMES:
Alveolar-arterial oxygen gradient (A-a DO2) | one hour of exposure to treatment gas
oxygen saturation by pulse oximetry (SpO2) | continuously through the study
need for mechanical ventilation | Continuously through the study
duration of oxygen therapy | continuously through the study
Methemoglobin level in post-ductal arterial blood (MetHb) | Hourly until completion of study in infant
Platelet count | As needed if bleeding
Systemic blood pressure | hourly
Environmental NO and NO2 exposure | Hourly

CONTACTS AND LOCATIONS:
Overall Officials: Namasivayam Ambalavanan, MD, Principal Investigator — University of Alabama at Birmingham; Waldemar A Carlo, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Regional Neonatal ICU, University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] Ambalavanan N, St John E, Carlo WA, Bulger A, Philips JB 3rd. Feasibility of nitric oxide administration by oxygen hood in neonatal pulmonary hypertension. J Perinatol. 2002 Jan;22(1):50-6. doi: 10.1038/sj.jp.7210652. PMID 11840243